CLINICAL TRIAL: NCT02437422
Title: A Phase Ib, Open-Label, Single Arm Study to Assess the Safety, Pharmacokinetics, and Impact on Humoral Sensitization of SANGUINATE Infusion in Patients With End-Stage Renal Disease (ESRD)
Brief Title: Study to Assess the Safety and Impact on Humoral Sensitization of SANGUINATE in Patients With End Stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGTP-001
Record Dates: First submitted 2015-04-06; First posted 2015-05-07 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — PEGylated carboxyhemoglobin bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SANGUINATE (Experimental): Single infusion of SANGUINATE
  Interventions: Biological: SANGUINATE

INTERVENTIONS:
Biological: SANGUINATE — Single two-hour infusion of SANGUINATE
  Other Names: (pegylated carboxyhemoglobin bovine)

SUMMARY:
A Phase Ib, Open-Label, Single Arm Study to Assess the Safety, Pharmacokinetics, and Impact on Humoral Sensitization of SANGUINATE Infusion in Patients with End Stage Renal Disease (ESRD).

DETAILED DESCRIPTION:
The purpose of the study is to investigate the safety of SANGUINATE on humoral sensitization in End Stage Renal Disease (ESRD) patients receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with End State Renal Disease requiring renal replacement therapy.
2. Age 18 - 65 years of age who are on maintenance hemodialysis for at least 3 months prior to the study start;
3. Stable dialysis treatment regimen 3 times per week for ≥ 2 months prior to screening visit;
4. Hemoglobin >7.5 g/dL with or without clinical symptoms;
5. Women of childbearing potential must have a negative serum pregnancy test and must use a reliable method of contraception during the study period;
6. Signed and dated informed written consent by the subject or his/her legally authorized representative;

Exclusion Criteria:

1. In the judgment of the investigator the patient is not a good candidate for the study;
2. Blood transfusion with in the last 90 days from date of Screening;
3. Symptoms or electrocardiogram (ECG)-based signs of acute myocardial infarction, Unstable angina pectoris, decompensated heart failure, third degree heart block or cardiac arrhythmia associated with hemodynamic instability;
4. Total bilirubin greater than 1.5 mg/dL or transaminase (ALT, AST) elevations greater than 2 times the upper limit of the laboratory reference range or evidence of significant hepatic insufficiency;
5. Concurrent or prior treatment within 90 days of Screening with an investigational medication;
6. Chronic treatment (as determined by the Investigator) with any immunosuppressive medication (including corticosteroids) within the past 90 days of Screening;
7. Evidence or history of regular alcohol abuse;
8. Screening laboratory result(s) determined to be clinically significant by the investigator;
9. Screening laboratory result indicating HIV-positivity, or previously diagnosed with AIDS, AIDS related complex or any other immunodeficiency;
10. Screening laboratory result or laboratory results performed within one year indicating positivity for hepatitis B surface antigens, hepatitis B core antibodies, or hepatitis C antibodies;
11. Uncontrolled Diabetes Mellitus (Patients with HbA1c > 9% at screening)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2015-11-18 (Actual)

PRIMARY OUTCOMES:
Safety of study treatment as determined by changes in vital signs, electrocardiographic assessments, clinical signs, and bio-analytical measures (e.g., blood chemistry, hematology), and reported adverse events following infusion | 90 days
  Composite endpoint with multiple vital signs, ECGs, clinical assessments and bio-analytical lab measurements over the 90 day time frame.

SECONDARY OUTCOMES:
Mean change in the number of HLA-Antibody specificities determined by single antigen bead assays | 90 days
  Antibody testing Human leukocyte antigen- antibody (HLA-Ab) HLA Tissue Typing (screening visit only) Calculated Panel Reactive Antibody (CPRA)
Mean change in the overall strength of HLA-Antibody specificities determined by single antigen bead assays | 90 days
  Antibody testing Human leukocyte antigen- antibody (HLA-Ab) HLA Tissue Typing (screening visit only) Calculated Panel Reactive Antibody (CPRA)
Mean change in the calculated panel reactive antibody (CPRA) | 90 days
  Antibody testing
Percent of patients with an increase in number of HLA-Ab specificities determined by single antigen bead assays | 90 Days
  Antibody testing
Percent of patients with an increase in CPRA | 90 Days
  Antibody testing
Pharmacokinetic profile as determined from blood plasma over time (Tmax, Cmax, AUC, half-life, coefficient of variation, and the apparent elimination rate constant) | 22 Days
Percent of patients with an increase in the overall strength of HLA-Antibodies | 90 Days
  Antibody testing

CONTACTS AND LOCATIONS:
Overall Officials: Bassam G Abu Jadweh, MD, Principal Investigator — University of Cincinnati/ Division of Nephrology
Locations (1):
- University of Cincinnati/ Division of Nephrology, Cincinnati, Ohio, United States